CLINICAL TRIAL: NCT04503486
Title: Relationship Between Grip and Quadriceps Strength on Quality of Life in ICU Survivors
Brief Title: Relationship Between Muscle Strength and Quality of Life in ICU Survivors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Rousseau, head of clinic, University of Liege
Other Study IDs: MQV-USI
Record Dates: First submitted 2020-08-01; First posted 2020-08-07 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Critical Illness; Muscle Strength; Quadriceps Strength; Grip Strength; Quality of Life
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: handgrip strength — measure of handgrip strength using Jamar Dynamometer and a standardized protocol, strength expressed in kg
Diagnostic Test: quadriceps strength — maximal isometric quadriceps strength measured using a handheld dynamometer and a standardized protocol, strength expressed in Newton

SUMMARY:
The aim is to study the impact of muscle strength measured in ICU and after ICU discharge on health-related quality of life measured after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* critically ill patients with an ICU stay of at least 7 days
* collaborative

Exclusion Criteria:

* non collaborative, confusion, coma
* limb paresis or plegia
* patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the study includes patients in ICU after a stay of at least 7 days. They are included as soon as they are collaborative.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
health-related quality of life | 1 month after ICU discharge
  assessed using the Sarcopenia Quality of Life (SARQOL) questionnaire short form: 8 questions with qualitative responses
health-related quality of life | 3 months after ICU discharge
  assessed using the Sarcopenia Quality of Life (SARQOL) questionnaire short form: 8 questions with qualitative responses
health-related quality of life | 6 months after ICU discharge
  assessed using the Sarcopenia Quality of Life (SARQOL) questionnaire short form: 8 questions with qualitative responses
health-related quality of life | 1 month after ICU discharge
  assessed using the EuroQOL 5 dimensions (EQ-5D) questionnaire: a first part assess the 5 dimensions of health state (each dimension is scored from 1 to 3, 3 indicating extreme problems). A second part is visual analog scale ranging from 0 (the worst health you can imagine) to 100 (the best health you can imagine)
health-related quality of life | 3 months after ICU discharge
  assessed using the EuroQOL 5 dimensions (EQ-5D) questionnaire: a first part assess the 5 dimensions of health state (each dimension is scored from 1 to 3, 3 indicating extreme problems). A second part is visual analog scale ranging from 0 (the worst health you can imagine) to 100 (the best health you can imagine)
health-related quality of life | 6 months after ICU discharge
  assessed using the EuroQOL 5 dimensions (EQ-5D) questionnaire: a first part assess the 5 dimensions of health state (each dimension is scored from 1 to 3, 3 indicating extreme problems). A second part is visual analog scale ranging from 0 (the worst health you can imagine) to 100 (the best health you can imagine)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No